CLINICAL TRIAL: NCT04446728
Title: Implementation of Family Psychosocial Risk Assessment in Pediatric Cancer With The Psychosocial Assessment Tool (PAT)
Brief Title: Implementation of Family Psychosocial Risk Assessment in Pediatric Cancer
Acronym: PAT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Collaborators: Children's Hospital of Philadelphia (Other); American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Anne E Kazak, PhD, ABPP, Center Director, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AK001
Record Dates: First submitted 2020-06-02; First posted 2020-06-25 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Cancer
Keywords: Families; Psychosocial; Health equity
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Masking Description: This is an implementation trial in which institutions are assigned to conditions. There is no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strategy I.Training (Active Comparator): Sites randomized to Strategy I will receive a three hour training webinar in preparing for implementation of the PAT in their center.
  Interventions: Behavioral: Training Webinar
- Strategy II.Training+Implementation Enhanced Resources (TIER) (Active Comparator): Sites randomized to Strategy II will identify a Champion for screening and will participate in a monthly consultation call in addition to completing the three hour training webinar for implementing the PAT in their center.
  Interventions: Behavioral: Training Webinar; Behavioral: Training Webinar Plus Implementation Enhanced Resources (TIER)

INTERVENTIONS:
Behavioral: Training Webinar — The training webinar is a three hour training. The purpose of the study is to implement the Psychosocial Assessment Tool (PAT) in their center.
Behavioral: Training Webinar Plus Implementation Enhanced Resources (TIER) — In addition the Training Webinar, sites randomized to Strategy II will identify a Champion and will participate in monthly consultation calls in support of implementation of the PAT
  Arms: Strategy II.Training+Implementation Enhanced Resources (TIER)

SUMMARY:
The diagnosis and treatment of pediatric cancer adversely affects multiple levels of the social ecology, including patient and caregiver physical and psychosocial health. It is the strong recommendation from the first Standard of the Psychosocial Standards of Care in Pediatric Cancer that cancer centers engage in universal, systematic, psychosocial risk screening for newly diagnosed patients and their families. Universal screening at diagnosis fosters early identification of psychosocial risks and provides the opportunity to match psychosocial care to the level of family need for more equitable, effective and integrated services. However, few programs offer such care in an efficient, comprehensive, and consistent manner, potentially resulting in insufficient care that magnifies inequities in outcomes. To support pediatric cancer centers in their goal of meeting the first Standard of Psychosocial Care, this study will compare two implementation strategies for the Psychosocial Assessment Tool (PAT), a validated parent report screener of family psychosocial risk in English and Spanish, in a cluster randomized trial across 18 pediatric cancer programs in the United States.

DETAILED DESCRIPTION:
Background: Childhood cancer affects multiple levels of the social ecology, including social determinants of health (e.g. financial and resource issues, child and family problems). The 2015 Standards of Psychosocial Care in Pediatric Cancer outline optimal psychosocial care, starting with a standard devoted to assessment of psychosocial healthcare needs. The Psychosocial Assessment Tool (PAT) is a validated family psychosocial risk screener now ready for broad implementation. Method: The PAT will be implemented across a national sample of 18 pediatric cancer programs in a comparative effectiveness study, guided by the Interactive Systems Framework for Dissemination and Implementation, comparing two Strategies. It is hypothesized that implementation will be more successful at the patient/family, provider, and institutional level when Training (Strategy I) is combined with Implementation Expanded Resources (Strategy II). The trial will be informed by input from Stakeholders and will result in a web-based Toolkit for dissemination nationally. Sites will be randomized to cohort (one of three years) and strategy (Strategy I, II) for the trial. Outcomes include adoption and penetration of screening (patient/family), staff job satisfaction/burnout (provider), and cost effective use of resources consistent with family risk (institution). Discussion Use of the PAT across children's cancer programs nationally can achieve the assessment Standard and deliver psychosocial care matched to family need for all patients, especially those most impacted by health inequities.

Based on the Interactive Systems Framework for Dissemination and Implementation (ISF), this study is a comparative effectiveness trial of the two strategies at 18 childhood cancer centers of three sizes based on new patients per year, examining family (penetration, health equity), provider (feasibility, acceptability, burnout and job satisfaction), and institution (adoption, sustainability, costs) implementation outcomes.7 Sites will be randomized to time of implementation (three cohorts) and Strategy (two - I, II).

Aim. Compare the two theoretically based and empirically informed strategies to implement the PAT in English and Spanish using a cluster randomized controlled trial. Compared to Training:

H1. At the patient/family level, TIER will be associated with: a) a higher proportion of families of newly diagnosed children screened and provided with feedback (penetration); and b) higher rates of screening for ethnic minority and socioeconomically diverse families (health equity).

H2. At the provider level, TIER will be: a) more feasible and rated as appropriate and acceptable; b) associated with greater engagement in addressing health disparities; and c) associated with less burnout and better job satisfaction.

H3. At the institution level, TIER will be associated with: a) a higher rate of site participation (adoption), b) more positive perceptions of implementation benefits and fewer challenges (sustainability); and c) psychosocial care better matched to need demonstrating a more equitable distribution of services and costs of care.

All sites, regardless of randomization to Strategy I or II, will participate in a 3-hour professionally prepared internet based learning session (webinar) at the beginning of their cohort. Each site PI, all staff who will be directly involved in screening, and the research coordinator will participate. For sites randomized to Strategy II, the Champion will also attend. The investigators will work with sites to identify the team that will participate in screening and the Champion (in TIER) ("individuals who dedicate themselves to supporting, marketing, and driving through an implementation, overcoming indifference or resistance that the intervention may encounter in an organization"), recognizing that these determinations will vary across programs. The webinar will be professionally prepared to be engaging and effective as an educational approach with resource materials provided (Develop Educational Materials, Distribute Educational Materials).

The training webinar will include all information necessary to access the web-based PAT. Sites will be provided with a User Agreement, user manual, and access to the password protected site. The completed PAT is scored immediately and a summary of the score and clinical concerns identified is sent. Only de-identified data will be transmitted to the study data core. Sites will be supported in the technical aspects of the implementation related to using the web-based forms (Centralize Technical Assistance). If any pattern of problems with technical aspects of implementation is identified, the study staff will communicate with sites promptly. During training, each site PI and staff involved in screening will develop a specific implementation plan, describing who will implement the PAT, who will be screened, where results will be stored, how results will be communicated and how results will be used (Develop a Formal Implementation Blueprint). For TIER, the Plan includes questions about the Champion and the Consultation Calls.

Strategy I. For sites randomized to Strategy I (Training), the webinar is the implementation condition. Sites will also receive technology support, as needed, throughout the one-year implementation period. These strategies correspond to implementation strategies: creating a structure for implementation including creating implementation teams, developing an implementation plan.2

Strategy II. Strategy II, Training + Implementation Expanded Resources (TIER), includes the same webinar and technical support as in Strategy I with the addition of two evidence-based resources that may improve implementation (as finalized from analysis of Aim 1 interviews). The Site PI and center staff conducting screening will participate in a monthly one-hour PAT Implementation Consultation Call (Provide Ongoing Consultation, Create a Learning Collaborative). The group format of this strategy is intended to foster group problem-solving about common issues in implementation and provide peer support for those implementing the PAT. The data regarding implementation progress and challenges from the calls will be addressed in subsequent calls and will be considered in the development of the Toolkit. Second, sites will identify a Champion for PAT implementation (Identify and Prepare Champions), most likely be a division chief, nurse in a leadership role, or clinical administrator.

At the Patient/Family level the following data for the English and Spanish versions of the PAT will be reported monthly: new patients meeting eligibility requirements as outlined on the PAT Implementation Plan (n); patients with documentation of PAT screening (n); patients with evidence of family feedback letter (n); demographic data (race, ethnicity, zip code, insurance). As part of the PAT Implementation Plan, the Site PI and Coordinator will determine institution-specific ways to identify new patients and their demographic characteristics.

At the Provider level the Site PI and staff identified as screeners will complete self-report measures at baseline and at 6 and 12 months.

There are four outcomes at the Institution level. The first outcome is adoption, or the intention of sites to use the PAT, by examining the site participation rate. To evaluate the extent to which screening is perceived as an asset to the institution electronic health record data (EHR) data will be extracted and aggregated at the site level for each family at 30, 60 and 90 days after screening. It provides a sum of hospital based services and external referrals and the number and length of inpatient and outpatient visits, missed appointments and evidence of non-adherence or difficulties in delivering care, allowing determination of healthcare utilization or medical services delivered. Cost will be assessed to understand the relationship among PAT risk level, psychosocial services provided, and aspects of medical care that may reflect unnecessary or inefficient services. Because the care provided may be related to the intensity of medical treatment, the Intensity of Treatment Scale will be used.

Analysis

H1. ANOVA will compare the effectiveness of the two implementation strategies on penetration and health equity. The outcomes are proportions: families screened/families eligible, families provided feedback/families screened, ethnic minority families screened/ethnic minority families eligible, low socioeconomic status (SES) families screened/low SES families eligible. Interclass Correlation Coefficients (ICC) among the clusters will be calculated and used to adjust for the cluster effect.

H2. Three sets of outcome variables - perception of implementation, engagement in addressing health disparities, and burnout/job satisfaction - will be tested. A two group analysis with the framework of Structural Equation Modeling (SEM) will be conducted to compare the effectiveness of the two strategies. To test the effect of time (T1, T2, T3), latent growth curve analysis will be conducted; it is expected that provider outcomes will improve over time. Analyses will be performed using Mplus 5.0 with ML estimation for outcome variables that meet the distribution assumptions, and with Robust Least Weighted Squares (WLSMV) estimation for outcome variables that do not. Potential mediating effects of favorable perception of implementation on provider job satisfaction and burnout will be examined using mediation models. TIER is expected to be associated with more favorable perceptions of implementation, which in turn will lead to less burnout and higher job satisfaction.

H3. At the institution level adoption of the PAT will be measured by a ratio of sites that initiate implementation/sites that agreed (H3a). If substitutions are necessary, sites that are newly invited will be added to the denominator and adoption calculated by total acceptances/total invited. ANOVA will be conducted to compare the effectiveness of the two strategies. For H3b sustainability (PIQ perceptions of implementation benefits and challenges), ANOVA will be conducted to compare the effectiveness of the two strategies on benefits and challenges. For H3c the interest is in the extent to which psychosocial care is matched to need and the extent to which intensive medical and psychosocial services are delivered for those most in need. There has not yet been established a cost-effectiveness threshold or criterion to which to compare costs of screening with these two implementation strategies, necessitating our consideration of valued outcomes in the psychosocial screening literature and resources available. ANOVA will be conducted to test whether psychosocial care is matched with levels of psychosocial risks, resulting in a 2 (Strategy) x 3 (psychosocial risks: clinical, targeted, universal) design on distribution of services and costs of care. It is expected that the 3 levels of the Pediatric Psychosocial Preventative Health Model (PPPHM) will be related to number and costs of services provided as measured on the Psychosocial Services and Medical Treatment Checklist (PSMTC). Additional analyses will be conducted to compare English speaking and Spanish speaking families, different ethnicity, race, and SES and insurance status on the outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* Sites were selected in advance based on data collected in a previous study regarding psychosocial staffing in the pediatric cancer program.
* Sites that were at or above the median for size of their psychosocial staff were eligible. - --
* Site selection took into consideration number of new pediatric cancer patients annually, geographical representation and sites with significant proportions of Spanish speaking families and/or families of low socioeconomic status.

Exclusion Criteria:

- Sites with psychosocial staffing below the median in the prior study were not eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Families screened | At conclusion of cohort year (12 months post baseline)
  Number of families screened divided by number of families eligible
Site Participation Rate | At conclusion of the study (12 months post baseline)
  Number of sites that completed the study divided by sites enrolled
Families provided feedback | At conclusion of cohort year (12 months post baseline)
  Number of families provided feedback divided by number of families screened
Ethnic minority families screened | At conclusion of cohort year (12 months post baseline)
  Number of ethnic minority families screened divided by number of ethnic minority families eligible
Physician Engagement in Addressing Racial and Ethnic Health Care Disparities (AREA) scale | Baseline, 6 and 12 months
  Changes in level of engagement in addressing health disparities as measured by the AREA, a 9 point scale with a 5 point likert response. Total scores range from 0 to 36 with higher scores indicating higher level of engagement
Maslach Burnout Inventory (MBI) | Baseline, 6 and 12 months
  Changes in burnout measured with this 22 item scale with a items on a 7 point Likert scale, higher scores indicate higher job satisfaction. Range of scores is from 0 to 42.
Acceptability of Intervention Measure (AIM) | Baseline, 6 months, 12 months
  Changes in acceptability of the PAT using this four item survey on a 5 point likert scale; range of scores is from 5 to 25; higher score is higher acceptability
Intervention Appropriateness Measure (IAM) | Baseline, 6 months, 12 months
  Changes in perceived appropriateness of the PAT using this four item survey on a 5 point likert scale; range of scores is from 5 to 25; higher score is higher appropriateness
Feasibility of Intervention Measure (FIM) | Baseline, 6 months, 12 months
  Changes in perceptions of the feasibility of using the PAT measured with this four item survey on a 5 point likert scale; range of scores is from 5 to 25; higher score is higher feasibility

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Children's Health, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share de-identified data upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At conclusion of study
Access Criteria: Data sharing will be considered with clinical leaders, investigators, policy makers and cancer advocates interested in implementation strategies for psychosocial screening and care.

REFERENCES:
- [Derived] Deatrick JA, Kazak AE, Scialla MA, Madden RE, McDonnell GA, Okonak K, Barakat LP. Advancing health equity in pediatric cancer through implementation of universal family psychosocial risk screening. Psychooncology. 2022 Sep;31(9):1483-1490. doi: 10.1002/pon.5978. Epub 2022 Jul 1. PMID 35726382
- [Derived] Deatrick JA, Kazak AE, Madden RE, McDonnell GA, Okonak K, Scialla MA, Barakat LP. Using qualitative and participatory methods to refine implementation strategies: universal family psychosocial screening in pediatric cancer. Implement Sci Commun. 2021 Jun 5;2(1):62. doi: 10.1186/s43058-021-00163-4. PMID 34090525
- [Derived] Kazak AE, Deatrick JA, Scialla MA, Sandler E, Madden RE, Barakat LP. Implementation of family psychosocial risk assessment in pediatric cancer with the Psychosocial Assessment Tool (PAT): study protocol for a cluster-randomized comparative effectiveness trial. Implement Sci. 2020 Jul 29;15(1):60. doi: 10.1186/s13012-020-01023-w. PMID 32727493